CLINICAL TRIAL: NCT03786432
Title: A Prospective Clinical Pilot Study Of Fusion Rates Using Spira™-C Titanium 3-D Printed Interbody Device For Anterior Cervical Discectomy And Fusion
Brief Title: Prospective Study of Fusion Rates Using Spira-C Device for Anterior Cervical Discectomy and Fusion Surgery
Acronym: ACDF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Could not continue enrollment due to discontinuation of funding
Sponsor: Corewell Health East (Other)
Collaborators: Camber Spine Technologies (Industry)
Responsible Party: Principal Investigator, Jad Khalil MD, Orthopaedic Spine surgeon and Assistant Professor of Orthopaedic Surgery, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-378
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Cervical Radiculopathy; Cervical Disc Disease
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Spira-C Interbody Device (Experimental): 40 subjects undergoing anterior cervical discectomy and fusion surgery using Spira-C titanium interbody device
  Interventions: Device: Spira-C Interbody Device

INTERVENTIONS:
Device: Spira-C Interbody Device — 40 subjects undergoing anterior cervical discectomy and fusion surgery using Spira-C titanium interbody device

SUMMARY:
The objective of this study is to perform a prospective, single-arm clinical evaluation utilizing the Spira™-C 3-D printed titanium interbody device for treatment of degenerative disc disease and spinal stenosis of the cervical spine to evaluate fusion status and patient reported outcomes. The primary objective is fusion status or bony healing within the device. Patient reported outcomes, i.e. pain, function, and quality of life will also be measured postoperatively.

DETAILED DESCRIPTION:
This is a post-market, single-arm, prospective clinical study to evaluate fusion status and patient reported outcomes using the Spira-C titanium interbody cage for degenerative disc disease where single-level ACDF surgery is indicated. The treatment group will consist of 40 subjects treated with the Spira™-C interbody device at one level. Patients with a diagnosis of cervical degenerative disc disease and/or spinal stenosis, radiculopathy or myelopathy and planning to undergo a 1-level ACDF surgery between C3-C7 will be screened and consented, if eligibility requirements are met. Once the subject has been enrolled and the surgery has taken place; data will be collected regarding the surgical details will be collected. Subjects will be followed up postoperatively at 6-weeks, 3-months, 6-months, and 12-months as per standard of care, at the private practice or clinic. Subjects will be asked to complete questionnaires regarding pain, function, and quality of life before and after surgery during the postoperative follow-up visits. Radiographic assessments will be performed at all postoperative visits; fusion status will be measured using cervical x-rays and CT scan at 12 months. Radiographs will also be utilized to assess for device-related complications, including implant failure. Any clinically significant complications related to the device will be recorded as an adverse event. This study design reflects the current standard of care for cervical degenerative disc disease and spinal stenosis with symptoms of radiculopathy or myelopathy. Data collected from subjects treated with the Spira™-C Interbody Device will be compared to historical data based on literature review of polyetheretherketone (PEEK) cage fusion rates and patient reported outcomes. Anterior cervical discectomy and fusion using an interbody device with plate and screw fixation is the treatment of choice after conservative therapies (non-surgical, i.e., physical therapy, epidural steroid injections, pain medications) have been exhausted.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age and skeletally mature
2. Able to provide consent
3. Undergoing a primary, single-level ACDF between C3-C7
4. Diagnosis of symptomatic degenerative disc disease
5. Neck pain and/or radicular symptoms with a baseline Visual Analog Scale score of ≥ 4cm (0-10cm scale)
6. Baseline Neck Disability Index score of ≥ 20
7. Attempted at least 6-weeks of conservative non-operative treatment

Exclusion Criteria:

1. Any prior history of cervical fusion
2. Requires cervical fusion of more than one level
3. Acute cervical spine trauma requiring immediate intervention
4. BMI > 40
5. Active systemic bacterial or fungal infection or infection at the operative site
6. History of vertebral fracture or osteoporotic fracture
7. Current treatment with chemotherapy, radiation, immunosuppression or chronic steroid therapy
8. History of osteoporosis, osteopenia, or osteomalacia that would contraindicate spinal surgery
9. Psychological or physical condition in the opinion of the investigator that would interfere with completing study participation including completion of patient reported outcomes
10. History of neurological condition in the opinion of the investigator that may affect cervical spine function and pain assessments
11. Subjects with a history of cancer must be disease free for at least 3 years; with the exception of squamous cell skin carcinoma
12. Pregnant, or plans on becoming pregnant
13. History of allergy to titanium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jad G Khalil, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGilvray KC, Easley J, Seim HB, Regan D, Berven SH, Hsu WK, Mroz TE, Puttlitz CM. Bony ingrowth potential of 3D-printed porous titanium alloy: a direct comparison of interbody cage materials in an in vivo ovine lumbar fusion model. Spine J. 2018 Jul;18(7):1250-1260. doi: 10.1016/j.spinee.2018.02.018. Epub 2018 Feb 26. PMID 29496624
- [Background] Li ZJ, Wang Y, Xu GJ, Tian P. Is PEEK cage better than titanium cage in anterior cervical discectomy and fusion surgery? A meta-analysis. BMC Musculoskelet Disord. 2016 Sep 1;17(1):379. doi: 10.1186/s12891-016-1234-1. PMID 27585553
- [Background] Cabraja M, Oezdemir S, Koeppen D, Kroppenstedt S. Anterior cervical discectomy and fusion: comparison of titanium and polyetheretherketone cages. BMC Musculoskelet Disord. 2012 Sep 14;13:172. doi: 10.1186/1471-2474-13-172. PMID 22978810
- [Background] Rao PJ, Pelletier MH, Walsh WR, Mobbs RJ. Spine interbody implants: material selection and modification, functionalization and bioactivation of surfaces to improve osseointegration. Orthop Surg. 2014 May;6(2):81-9. doi: 10.1111/os.12098. PMID 24890288
- [Background] Hsu MR, Haleem MS, Hsu W. 3D Printing Applications in Minimally Invasive Spine Surgery. Minim Invasive Surg. 2018 Apr 1;2018:4760769. doi: 10.1155/2018/4760769. eCollection 2018. PMID 29805806
- [Background] Niu CC, Liao JC, Chen WJ, Chen LH. Outcomes of interbody fusion cages used in 1 and 2-levels anterior cervical discectomy and fusion: titanium cages versus polyetheretherketone (PEEK) cages. J Spinal Disord Tech. 2010 Jul;23(5):310-6. doi: 10.1097/BSD.0b013e3181af3a84. PMID 20124907
- [Background] Lee YS, Kim YB, Park SW. Risk factors for postoperative subsidence of single-level anterior cervical discectomy and fusion: the significance of the preoperative cervical alignment. Spine (Phila Pa 1976). 2014 Jul 15;39(16):1280-7. doi: 10.1097/BRS.0000000000000400. PMID 24827519
- [Background] Chen Y, Wang X, Lu X, Yang L, Yang H, Yuan W, Chen D. Comparison of titanium and polyetheretherketone (PEEK) cages in the surgical treatment of multilevel cervical spondylotic myelopathy: a prospective, randomized, control study with over 7-year follow-up. Eur Spine J. 2013 Jul;22(7):1539-46. doi: 10.1007/s00586-013-2772-y. Epub 2013 Apr 9. PMID 23568254
- [Background] Seaman S, Kerezoudis P, Bydon M, Torner JC, Hitchon PW. Titanium vs. polyetheretherketone (PEEK) interbody fusion: Meta-analysis and review of the literature. J Clin Neurosci. 2017 Oct;44:23-29. doi: 10.1016/j.jocn.2017.06.062. Epub 2017 Jul 21. PMID 28736113
- [Background] Wilcox B, Mobbs RJ, Wu AM, Phan K. Systematic review of 3D printing in spinal surgery: the current state of play. J Spine Surg. 2017 Sep;3(3):433-443. doi: 10.21037/jss.2017.09.01. PMID 29057355

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a single-arm, post market study to evaluate fusion status and patient reported outcomes using the FDA approved Spira-C Titanium Interbody Device at one level. Patients with a diagnosis of cervical degenerative disc disease and/or spinal stenosis, radiculopathy or myelopathy and planning to undergo a 1-level ACDF surgery between C3-C7 were screened and enrolled in the study.
Period: Overall Study
Arm/Group | Spira-C Interbody Device
Started | 13
Completed 12 Month Visit | 8
Completed 12 Month CT Scan | 7
Completed | 7
Not Completed | 6
Not completed — Screen Failure after consent | 1
Not completed — Lost to Follow-up | 4
Not completed — did not complete 12 month CT scan | 1

BASELINE CHARACTERISTICS:
Population: Demographics not collected for 1 participants who was a screen failure.
Groups:
- Spira-C Interbody Device: subjects undergoing anterior cervical discectomy and fusion surgery using Spira-C titanium interbody device
  Spira-C Interbody Device: subjects undergoing anterior cervical discectomy and fusion surgery using Spira-C titanium interbody device
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: Age in years] | 53 [39 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Successful Cervical Fusion Measured Radiographically
Description: Count of participants with successful cervical fusion as measured by CT scan and flexion/extension x-rays at 12-months as evidenced by the following three criteria: bony bridging, no development of pseudoarthrosis, and no presence of radiolucency at the treated cervical level
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up, 1 did not complete CT scan and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 7
Participants | 6

2. Secondary Outcome: Decreased Visual Analog Scale for Neck Pain
Description: Count of participants with equal to or greater than a 2-point decrease in patient reported outcomes as measured by Visual Analog Scale for pain (0-10 point scale, 0 = no pain and 10 = severe amount of pain) from baseline to 12-months in the neck region.
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 8
Participants | 6

3. Secondary Outcome: Decreased Neck Disability Index for Pain and Function
Description: Count of participants with equal to or greater than a 15-point decrease in patient reported outcomes as measured by Neck Disability Index (0-100 point scale, 0 = least amount disability, 100 = most severe disability) from baseline to 12-months.
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 8
Participants | 6

4. Secondary Outcome: Increased Quality of Life Measured by Short Form Health Survey-36 (SF-36)
Description: Count of participants with Equal to or greater than 15-point increase in patient reported general health score as measured by SF-36 (0-100 point scale, 0 = low favorable health state and 100 = most favorable health state) from baseline to 12-months.
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 8
Participants | 3

5. Secondary Outcome: Eating Assessment Tool-10 for Dysphagia
Description: Count of participants with score of less than 3 or equal to baseline in patient reported outcomes as measured by Eating Assessment Tool-10 from baseline to 12-months.
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 8
Participants | 7

6. Secondary Outcome: Worsening Neurological Deficit Per Cervical Spine Examination
Description: Count of participants with new or worsening neurological cervical spine deficit as evaluated by cervical spine (motor and sensory) examination from baseline to 12-months.
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up, 1 did not complete CT scan and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 7
Participants | 6

7. Secondary Outcome: Count of Participants With Revision Surgery by Month 12
Description: Count of participants with revision surgery by month 12
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 8
Participants | 0

8. Secondary Outcome: Count of Participants With Development of Pseudoarthrosis by Month 12
Description: Count of participants with development of pseudoarthrosis by month 12
Time Frame: 12 months postoperative
Population: 4 were lost to follow-up, 1 did not complete CT scan and 1 screen failure-no data out of 13 enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Spira-C Interbody Device
Number analyzed (Participants) | 7
Participants | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Spira-C Interbody Device
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of participants analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/32/NCT03786432/Prot_SAP_000.pdf